CLINICAL TRIAL: NCT01438203
Title: Early Use of Thrust Manipulation Versus Non-Thrust Manipulation: A Randomized Clinical Trial
Brief Title: Thrust Manipulation Versus Non-Thrust Manipulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walsh University (Other)
Responsible Party: Principal Investigator, Chad Cook, Principal Investigator, Walsh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Walsh 10-24
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Mechanical Low Back Pain
Keywords: manipulation; mobilization; low back pain; treatment
MeSH Terms: conditions — Low Back Pain | interventions — Mob protein, Bacteria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrust manipulation (Experimental): Clinicians will use thrust manipulation at a targeted level to provide the treatment on selected individuals
  Interventions: Procedure: Thrust manipulation
- Non-thrust manipulation (Active Comparator): Clinicians will apply non-thrust manipulation (targeted) as performed in a clinical manner for treatment for included individuals
  Interventions: Procedure: Non-thrust manipulation

INTERVENTIONS:
Procedure: Thrust manipulation — Thrust manipulation is a passive procedure which involves a high velocity low amplitude thrust to the spinal region
  Other Names: Manipualtion (Manip)
  Arms: Thrust manipulation
Procedure: Non-thrust manipulation — Non-thrust manipulation involves a low amplitude, low speed mobilization to the targeted region while adjusting the procedure based on patient feedback
  Other Names: Mobilization (Mob)
  Arms: Non-thrust manipulation

SUMMARY:
The objective of this study is to investigate the comparative benefit of thrust and non-thrust manipulation on a population of patients with low back pain. The investigators hypothesize that there will be no difference in 4 week outcomes or greater, between the two groups.

DETAILED DESCRIPTION:
Thrust manipulation is considered traditional spinal manipulation. Nonthrust manipulation is considered mobilization. The mobilization will be used in a similar manner as in clinical practice and this differs from past studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients, age 18 and older, with mechanically producible low back pain, who attend care at a physical therapy outpatient setting, will be screened for eligibility for the study.
* For patients to meet inclusion requirements, they had to display a within session change in pain and/or range of motion during the assessment phase of the clinical examination. In other words, as the clinician performed their assessment and applied a passive accessory assessment technique, the pain and/or range of motion improved during that session, which suggests a favorable outcome using a comparable treatment technique. This is hallmark clinical finding in the patient response model and has been proposed as both a predictor of a positive outcome and as a prognostic variable toward long-term improvements in impairments.

Exclusion Criteria:

* The presence of any red flags (i.e., tumor, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
* Signs consistent with nerve root compression (reproduction of low back or leg pain with straight leg raise at less than 45°
* Muscle weakness involving a major muscle group of the lower extremity,
* Diminished lower extremity muscle stretch reflex
* Diminished or absent sensation to pinprick in any lower extremity dermatome)
* Other exclusion criteria included prior surgery to the lumbar spine and current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | Baseline to discharge from therapy services (up to 4 months). An expected average is 4 weeks.
  Change score

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline to discharge from therapy services (up to 4 months). An expected average is 4 weeks.
  Change score

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Cook, PhD, Principal Investigator — Walsh University
Locations (1):
- Walsh University, North Canton, Ohio, United States

REFERENCES:
- [Derived] Cook CE, Learman KE, O'Halloran BJ, Showalter CR, Kabbaz VJ, Goode AP, Wright AA. Which prognostic factors for low back pain are generic predictors of outcome across a range of recovery domains? Phys Ther. 2013 Jan;93(1):32-40. doi: 10.2522/ptj.20120216. Epub 2012 Aug 9. PMID 22879443